CLINICAL TRIAL: NCT03972150
Title: An Open Label, Phase I Study of BI 836880 Monotherapy and Combination Therapy of BI 836880 and BI 754091 in Japanese Patients With Advanced Solid Tumours
Brief Title: A Study to Find the Best Dose of BI 836880 Alone and in Combination With BI 754091 in Japanese Patients With Different Types of Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1336-0012
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Results first posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1: 360 mg BI 836880 (Experimental): Patients with advanced solid tumors were administered intravenously (i.v.) 360 milligram (mg) of BI 836880 solution for infusion on Day 1 of each 3-week cycle until progressive disease, unacceptable toxicity, or other withdrawal criteria were met (Part 1).
  Interventions: Drug: BI 836880
- Part 1: 720 mg BI 836880 (Experimental): Patients with advanced solid tumors were administered intravenously (i. v.) 720 milligram (mg) of BI 836880 solution for infusion on Day 1 of each 3-week cycle until progressive disease, unacceptable toxicity, or other withdrawal criteria were met (Part 1).
  Interventions: Drug: BI 836880
- Part 2: 120 mg of BI 836880/ 240 mg Ezabenlimab (Experimental): Patients with advanced solid tumors were administered intravenously (i. v.) 120 milligram (mg) of BI 836880 solution for infusion and 240 mg Ezabenlimab (BI 754091) solution for infusion on Day 1 of each 3-week cycle until progressive disease, unacceptable toxicity, or other withdrawal criteria were met (Part 2). Part 2 commenced after completion of Part 1.
  Interventions: Drug: BI 836880; Drug: BI 754091
- Part 2: 360 mg BI 836880/ 240 mg Ezabenlimab (Experimental): Patients with advanced solid tumors were administered intravenously (i. v.) 360 milligram (mg) of BI 836880 solution for infusion and 240 mg Ezabenlimab (BI 754091) solution for infusion on Day 1 of each 3-week cycle until progressive disease, unacceptable toxicity, or other withdrawal criteria were met (Part 2). Part 2 commenced after completion of Part 1.
  Interventions: Drug: BI 836880; Drug: BI 754091
- Part 2: 720 mg BI 836880 / 240 mg Ezabenlimab (Experimental): Patients with advanced solid tumors were administered intravenously (i. v.) 720 milligram (mg) of BI 836880 solution for infusion and 240 mg Ezabenlimab (BI 754091) solution for infusion on Day 1 of each 3-week cycle until progressive disease, unacceptable toxicity, or other withdrawal criteria were met (Part 2). Part 2 commenced after completion of Part 1.
  Interventions: Drug: BI 836880; Drug: BI 754091

INTERVENTIONS:
Drug: BI 836880 — Solution for infusion
Drug: BI 754091 — Solution for infusion
  Arms: Part 2: 120 mg of BI 836880/ 240 mg Ezabenlimab; Part 2: 360 mg BI 836880/ 240 mg Ezabenlimab; Part 2: 720 mg BI 836880 / 240 mg Ezabenlimab

SUMMARY:
The primary objective of this trial is:

Part I

* To determine Maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of BI 836880 monotherapy Part II
* To determine MTD and/or RP2D of the combination therapy of BI 836880 and BI 754091

The secondary objectives are:

Part I

* To document the safety and tolerability, and characterise pharmacokinetics (PK) of BI 836880 as monotherapy Part II
* To document the safety and tolerability, and characterise PK of the combination therapy of BI 836880 and BI 754091

ELIGIBILITY:
Inclusion Criteria:

* Of legal age (according to local legislation) at screening. No upper limit.
* Signed and dated written informed consent in accordance with International Council on Harmonisation (ICH) Good Clinical Practice (GCP) and local legislation prior to admission to the trial.
* Male or female patients. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly, starting with the screening visit and through 6 months after the last dose of study treatment. A list of contraception methods meeting these criteria is provided in the patient information. The requirement of contraception does not apply to women of no childbearing potential and men not able to father a child, but they must have an evidence of such at screening.
* Patients with a confirmed diagnosis of advanced, unresectable, and/or metastatic solid tumours (any type). Measurable lesion not mandatory for participation in this trial.
* Patients with no therapy of proven efficacy, or who are not amenable to standard therapies.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
* Recovery from all reversible adverse events of previous anti-cancer therapies to baseline or Common Terminology Criteria for Adverse Events (CTCAE) grade 1, except for alopecia (any grade), sensory peripheral neuropathy, must be ≤ CTCAE grade 2 or considered not clinically significant.
* Adequate organ function.
* Further inclusion criteria apply.

Exclusion criteria:

* Known hypersensitivity to the trial drugs or their excipients or risk of allergic of anaphylactic reaction to drug product according to Investigator judgement (e.g. patient with history of anaphylactic reaction or autoimmune disease that is not controlled by nonsteroidal anti-inflammatory drugs (NSAIDs), inhaled corticosteroids, or the equivalent of ≤10 mg/day prednisone).
* Known history of human immunodeficiency virus (HIV) infection. Test results obtained in routine diagnostics are acceptable if done within 14 days before the informed consent date.
* Any of the following laboratory evidence of hepatitis virus infection.

  * Positive results of hepatitis B surface (HBs) antigen
  * Presence of hepatitis B core (HBc) antibody together with hepatitis virus B (HBV) Deoxyribonucleic acid (DNA)
  * Presence of hepatitis virus C (HCV) Ribonucleic acid (RNA) Test results obtained in routine diagnostics are acceptable if done within 14 days before the informed consent date.
* History of severe known hypersensitivity reactions to other mAbs.
* Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 4 weeks prior to the first dose of trial medication.
* Any investigational or anti-tumour treatment within 4 weeks or 5 half-life periods (whichever is shorter) prior to the initiation of trial treatment.
* Serious concomitant disease, especially those affecting compliance with trial requirements or which are considered relevant for the evaluation of the endpoints of the trial drug, such as neurologic, psychiatric, infectious disease or active ulcers (gastrointestinal tract, skin) or laboratory abnormality that may increase the risk associated with trial participation or trial drug administration, and in the judgment of the investigator would make the patient inappropriate for entry into the trial.
* Major injuries and/or surgery or bone fracture within 4 weeks of start of treatment, or planned surgical procedures during the trial period.
* Patients with personal or family history of QT prolongation and/or long QT syndrome, or prolonged QTcF (Corrected QT interval by Fridericia) at screening (>470 ms).
* Significant cardiovascular/cerebrovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of infarction within past 6 months, congestive heart failure >NYHA [New York Heart Association] class II).

Uncontrolled hypertension is defined as follows: Blood pressure in rested and relaxed condition ≥140 mmHg, systolic or ≥90 mmHg diastolic (with or without medication)

* Left Ventricular Ejection Fraction (LVEF) <50% measured locally by echocardiography
* History of severe haemorrhagic or thromboembolic event in the past 12 months (excluding central venous catheter thrombosis and peripheral deep vein thrombosis).
* Known inherited predisposition to bleeding or to thrombosis in the opinion of the investigator.
* Untreated brain metastasis(es) that may be considered active. Patients with previously treated brain metastases may participate provided they are stable (i.e., without evidence of progressive disease (PD) by imaging for at least 4 weeks prior to the first dose of trial treatment, and any neurologic symptoms have returned to baseline), and there is no evidence of new or enlarging brain metastases
* Patients who require full-dose anticoagulation (according to local guidelines). No Vitamin K antagonist and other anticoagulation allowed; Low Molecular Weight Heparin (LMWH) allowed only for prevention not for curative treatment.
* History (including current) of interstitial lung disease or pneumonitis within the last 5 years.
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Patients not expected to comply with the protocol requirements or not expected to complete the trial as scheduled. (e.g. chronic alcohol or drug abuse or any other condition that, in the investigator's opinion, makes the patient an unreliable trial participant).
* Patients who were previously treated in this trial.
* Patients with haematological malignancies.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial. Female patients of childbearing potential must have a negative urine or serum pregnancy test within 3 days prior to taking study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The serum pregnancy test must be negative for the patient to be eligible. Women who are nursing can be enrolled if they stop nursing. In this case, the patient cannot resume nursing even after discontinuation of study treatment.
* Further exclusion criteria apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2022-03-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Shizuoka Cancer Center, Shizuoka, Sunto-gun
  - National Cancer Center Hospital, Tokyo, Chuo-ku

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Yamamoto N, Koyama T, Shimizu T, Todaka A, Kawakami T, Erzen D, Sarashina A, Li B, Hou J, Yamazaki K. Phase I study of the VEGF/Ang-2 inhibitor BI 836880 alone or combined with the anti-programmed cell death protein-1 antibody ezabenlimab in Japanese patients with advanced solid tumors. Cancer Chemother Pharmacol. 2023 Jun;91(6):469-480. doi: 10.1007/s00280-023-04527-6. Epub 2023 May 4. PMID 37140602
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase I, open label, uncontrolled, non-randomized, two parts, dose-escalation design trial assessing the Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D), safety, tolerability, Pharmacokinetics (PK) and Pharmacodynamics (Pd) of BI 836880 monotherapy, and combination therapy of BI 836880 and BI 754091 in Japanese patients with different types of advanced cancer.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Part 1: 360 mg BI 836880 | Part 1: 720 mg BI 836880 | Part 2: 120 mg of BI 836880/ 240 mg Ezabenlimab | Part 2: 360 mg BI 836880/ 240 mg Ezabenlimab | Part 2: 720 mg BI 836880 / 240 mg Ezabenlimab
Started | 3 | 6 | 3 | 3 | 6
Completed | 0 | 0 | 0 | 1 | 3
Not Completed | 3 | 6 | 3 | 2 | 3
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0
Not completed — Progressive disease | 3 | 5 | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Treated set (TS) in monotherapy:
  This patient set included all patients enrolled in the trial who were documented to have administrated at least one dose of BI 836880 monotherapy.
  Treated set (TS) in combination therapy:
  This patient set included all patients enrolled in the trial who were documented to have administrated at least one dose of BI 836880 and ezabenlimab combination therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: 360 mg BI 836880 | Part 1: 720 mg BI 836880 | Part 2: 120 mg of BI 836880/ 240 mg Ezabenlimab | Part 2: 360 mg BI 836880/ 240 mg Ezabenlimab | Part 2: 720 mg BI 836880 / 240 mg Ezabenlimab | Total
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 6 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (15.7) | 54.8 (14.7) | 51.7 (12.0) | 57.3 (15.5) | 62.0 (8.8) | 57.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 1 | 4 | 13
  Male | 1 | 2 | 1 | 2 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 6 | 3 | 3 | 6 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 6 | 3 | 3 | 6 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of BI 836880 Monotherapy and Combination Therapy of BI 836880 and BI754091
Description: Maximum tolerated dose (MTD) of BI 836880 monotherapy (Part 1) and combination therapy of BI 836880 and BI75409 (Part 2). The MTD was defined as the highest dose with less than 25% risk of the true dose-limiting toxicity (DLT) rate being equal or above 0.33 (EWOC criterion) during the MTD evaluation period. The analysis of the MTD was based on a Bayesian logistic regression model (BLRM) guided by the escalation with overdose control principle. The estimated probability of a DLT at each dose level from the model was summarized using the following intervals:
  Underdosing: [0.00, 0.16) Targeted toxicity: [0.16, 0.33) Over toxicity: [0.33, 1.00]
Time Frame: First treatment cycle, the first 21 days following the start of trial medication.
Population: Dose escalation cohort treated set in monotherapy/combination therapy:
  This patients sets included all patients enrolled in dose escalation cohort of monotherapy/combination therapy who were documented to have administrated at least one dose of study medication and were evaluable for the MTD determination. This set is used for dose finding and MTD determination in Part I/Part II.
Measure: Number; unit: milligram
Groups:
- Part 1: Total BI 836880: Patients with advanced solid tumors were administered intravenously (i.v.) 360 milligram (mg) or 720 mg of BI 836880 solution for infusion on Day 1 of each 3-week cycle until progressive disease, unacceptable toxicity, or other withdrawal criteria were met (Part 1).
- Part 2: Total BI 836880/ 240 mg Ezabenlimab: Patients with advanced solid tumors were administered intravenously (i. v.) 120 milligram (mg) or 360 mg or 720 mg of BI 836880 solution for infusion and 240 mg Ezabenlimab (BI 754091) solution for infusion on Day 1 of each 3-week cycle until progressive disease, unacceptable toxicity, or other withdrawal criteria were met (Part 2). Part 2 commenced after completion of Part 1.
Arm/Group | Part 1: Total BI 836880 | Part 2: Total BI 836880/ 240 mg Ezabenlimab
Number analyzed (Participants) | 9 | 12
milligram | NA — Maximum tolerated dose was not reached as no DLTs were reported during the MTD evaluation period (Cycle 1) in Part 1. | NA — Maximum tolerated dose was not reached as no DLTs were reported during the MTD evaluation period (Cycle 1) in Part 2.

2. Primary Outcome: Number of Participants With Dose-limiting Toxicity (DLT) During the First Treatment Cycle
Description: Number of participants with DLT occurring during the first treatment cycle. DLT was defined as any of the following adverse events related to the treatment: Haematologic toxicities: -Any Grade 5 toxicity,-Neutropenia Grade 4 lasting for >7 days,-Grade ≥3 documented infection with neutropenia,-Febrile neutropenia (absolute neutrophil count <1.0 X 109 cells/L and fever ≥38.5C or a sustained temperature of ≥38.0 Centigrade (C) for more than 1 hour),-Grade 4 thrombocytopenia, or Grade 3 thrombocytopenia with bleeding,-Thrombocytopenia of any Grade which requires platelet transfusions,-Grade 4 anaemia unexplained by underlying disease,-Anaemia of any Grade which requires blood transfusions. Non-haematological toxicities: - Aspartate transaminase (AST) or Alanin-Aminotransferase (ALT) >3 times Upper Level of Normal (ULN) and concurrent total bilirubin >2 times ULN without initial findings of cholestasis,-≥ Grade 4 AST or ALT of any duration.
Time Frame: First treatment cycle, the first 21 days following the start of trial medication.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 360 mg BI 836880 | Part 1: 720 mg BI 836880 | Part 2: 120 mg of BI 836880/ 240 mg Ezabenlimab | Part 2: 360 mg BI 836880/ 240 mg Ezabenlimab | Part 2: 720 mg BI 836880 / 240 mg Ezabenlimab
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 6
Participants | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Maximum Measured Concentration of BI 836880 in Part 1 and Part 2 in Plasma (Cmax) at Cycle 1
Description: Maximum measured concentration of BI 836880 at Cycle 1 in Part 1 (monotherapy) and Part 2 (combination therapy) in plasma (Cmax) is reported.
Time Frame: Part 1(P1): Within 5 minutes(min) before, at 1 hour(h), 1.5h, 2.5h, 4.5h, 7.5h, 24h, 48h, 168h, 336h after Cycle 1 dose. Part 2(P2): Within 5 min before and at 1h, 2h15min, 6h, 24h, 168h, 336h after Cycle 1 dose. P1,P2: Within 5min before Cycle 2 dose.
Population: Pharmacokinetics parameter analysis set (PKS): The PK parameter analysis set (PKS) included all subjects from the Treated Set (TS) who provide at least one Pharmacokinetics (PK) parameter that was not excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram / milliliter (µg/mL)
Arm/Group | Part 1: 360 mg BI 836880 | Part 1: 720 mg BI 836880 | Part 2: 120 mg of BI 836880/ 240 mg Ezabenlimab | Part 2: 360 mg BI 836880/ 240 mg Ezabenlimab | Part 2: 720 mg BI 836880 / 240 mg Ezabenlimab
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 6
microgram / milliliter (µg/mL) | 131 (20.6) | 281 (22.7) | 50.4 (8.71) | 121 (21.6) | 316 (21.1)

4. Secondary Outcome: Area Under the Concentration-time Curve of BI 836880 in Part 1 and Part 2 in Plasma Over the Time Interval From 0 to 504 Hours (AUC0-504h) at Cycle 1
Description: Area under the concentration-time curve of BI 836880 in Part 1 (monotherapy) and in Part 2 (combination therapy) in plasma over the time interval from 0 to 504 hours (AUC0-504h) is reported.
Time Frame: Part 1(P1): Within 5 minutes(min) before and at 1 hour(h), 1.5h, 2.5h, 4.5h, 7.5h, 24h, 48h, 168h, 336h after Cycle 1 dose. Part 2(P2): Within 5min before and at 1h, 2h15min, 6h, 24h, 168h, 336h after Cycle 1 dose. P1,P2: Within 5min before Cycle 2 dose.
Population: PK parameter analysis set (PKS): The PK parameter analysis set (PKS) included all subjects from the Treated Set (TS) who provide at least one Pharmacokinetic (PK) parameter that was not excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter (h*µg/mL)
Arm/Group | Part 1: 360 mg BI 836880 | Part 1: 720 mg BI 836880 | Part 2: 120 mg of BI 836880/ 240 mg Ezabenlimab | Part 2: 360 mg BI 836880/ 240 mg Ezabenlimab | Part 2: 720 mg BI 836880 / 240 mg Ezabenlimab
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 6
hour*microgram/milliliter (h*µg/mL) | 22300 (24.4) | 50400 (24.5) | 8220 (7.68) | 21100 (28.5) | 50000 (24.3)

5. Secondary Outcome: Maximum Measured Concentration of BI 836880 in Part 1 in Plasma (Cmax) at Cycle 2
Description: Maximum measured concentration of BI 836880 at Cycle 2 in Part 1 (monotherapy) in plasma (Cmax) is reported.
Time Frame: Within 5 minutes (min) before and at 1 hour (h), 1.5h, 2.5h, 4.5h, 7.5h, 24h, 48h, 168h, 336h after dose in Cycle 2. Also, Within 5 min before Cycle 3 dose.
Population: Pharmacokinetics parameter analysis set (PKS): The PK parameter analysis set (PKS) included all subjects from the Treated Set (TS) who provide at least one PK parameter that was not excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram / milliliter (µg/mL)
Arm/Group | Part 1: 360 mg BI 836880 | Part 1: 720 mg BI 836880
Number analyzed (Participants) | 3 | 6
microgram / milliliter (µg/mL) | 178 (22.0) | 319 (24.0)

6. Secondary Outcome: Area Under the Concentration-time Curve of BI 836880 in Part 1 in Plasma Over the Time Interval From 0 to 504 Hours (AUC0-504h) at Cycle 2
Description: Area under the concentration-time curve of BI 836880 in Part 1 (monotherapy) at Cycle 2 in plasma over the time interval from 0 to 504 hours (AUC0-504h) is reported.
Time Frame: as for outcome 5
Population: PK parameter analysis set (PKS): The PK parameter analysis set (PKS) included all subjects from the Treated Set (TS) who provide at least one PK parameter that was not excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter (h*µg/mL)
Arm/Group | Part 1: 360 mg BI 836880 | Part 1: 720 mg BI 836880
Number analyzed (Participants) | 3 | 6
hour*microgram/milliliter (h*µg/mL) | 27600 (31.3) | 64900 (36.8)

7. Secondary Outcome: Maximum Measured Concentration of BI 836880 in Part 1 and Part 2 in Plasma (Cmax) at Cycle 4
Description: Maximum measured concentration of BI 836880 at Cycle 4 in Part 1 (monotherapy) and Part 2 (combination therapy) in plasma (Cmax) is reported.
Time Frame: Part 1(P1): Within 5 minutes (min) before and at 1 hour (h), 1.5h, 2.5h, 4.5h, 7.5h, 24h, 168h, 336h after Cycle 4 dose. Part 2(P2): Within 5min before and at 1 h, 2h15min, 6h, 24h, 168h, 336h after Cycle 4 dose. P1,P2: Within 5min before Cycle 5 dose.
Population: Pharmacokinetics parameter analysis set (PKS): The PK parameter analysis set (PKS) included all subjects from the Treated Set (TS) who provide at least one PK parameter that was not excluded. Only patients with no missing values are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram / milliliter (µg/mL)
Arm/Group | Part 1: 360 mg BI 836880 | Part 1: 720 mg BI 836880 | Part 2: 120 mg of BI 836880/ 240 mg Ezabenlimab | Part 2: 360 mg BI 836880/ 240 mg Ezabenlimab | Part 2: 720 mg BI 836880 / 240 mg Ezabenlimab
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 3
microgram / milliliter (µg/mL) | 184 (27.6) | 621 (6.83) | 55.9 (12.8) | 159 (31.6) | 398 (32.3)

8. Secondary Outcome: Area Under the Concentration-time Curve of BI 836880 in Part1 and Part 2 in Plasma Over the Time Interval From 0 to 504 Hours (AUC0-504h) at Cycle 4
Description: Area under the concentration-time curve of BI 836880 in Part 1 (monotherapy) and in Part 2 (combination therapy) at Cycle 4 in plasma over the time interval from 0 to 504 hours (AUC0-504h) is reported.
Time Frame: as for outcome 7
Population: PK parameter analysis set (PKS): The PK parameter analysis set (PKS) included all subjects from the Treated Set (TS) who provide at least one PK parameter that was not excluded. Only patients with no missing values are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter (h*µg/mL)
Arm/Group | Part 1: 360 mg BI 836880 | Part 1: 720 mg BI 836880 | Part 2: 120 mg of BI 836880/ 240 mg Ezabenlimab | Part 2: 360 mg BI 836880/ 240 mg Ezabenlimab | Part 2: 720 mg BI 836880 / 240 mg Ezabenlimab
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 3
hour*microgram/milliliter (h*µg/mL) | 35500 (46.6) | 122000 (14.2) | 10600 (6.81) | 31400 (37.4) | 79100 (16.4)

9. Secondary Outcome: Maximum Measured Concentration of Ezabenlimab (BI 754091) in Part 2 in Plasma (Cmax) at Cycle 1
Description: Maximum measured concentration of Ezabenlimab (BI 754091) at Cycle 1 in Part 2 (combination therapy) in plasma (Cmax) is reported.
Time Frame: Within 5 min before and at 1h, 2h15min, 6h, 24h, 168h, 336h after Cycle 1 dose. Also, Within 5 min before Cycle 2 dose.
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram / milliliter (µg/mL)
Arm/Group | Part 2: 120 mg of BI 836880/ 240 mg Ezabenlimab | Part 2: 360 mg BI 836880/ 240 mg Ezabenlimab | Part 2: 720 mg BI 836880 / 240 mg Ezabenlimab
Number analyzed (Participants) | 3 | 3 | 6
microgram / milliliter (µg/mL) | 83.9 (6.01) | 75.3 (25.4) | 104 (19.8)

10. Secondary Outcome: Area Under the Concentration-time Curve of Ezabenlimab (BI 754091) in Part 2 in Plasma Over the Time Interval From 0 to 504 Hours (AUC0-504h) at Cycle 1
Description: Area under the concentration-time curve of Ezabenlimab (BI 754091) in Part 2 (combination therapy) in plasma over the time interval from 0 to 504 hours (AUC0-504h) is reported.
Time Frame: Within 5 min before and at 1h, 2h15min, 6h, 24h, 168h, 336h after Cycle 1 dose. Also, Within 5 min before Cycle 2 dose.
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter (h*µg/mL)
Arm/Group | Part 2: 120 mg of BI 836880/ 240 mg Ezabenlimab | Part 2: 360 mg BI 836880/ 240 mg Ezabenlimab | Part 2: 720 mg BI 836880 / 240 mg Ezabenlimab
Number analyzed (Participants) | 3 | 3 | 6
hour*microgram/milliliter (h*µg/mL) | 18400 (5.28) | 15300 (23.8) | 16600 (26.4)

11. Secondary Outcome: Maximum Measured Concentration of Ezabenlimab (BI 754091) in Part 2 in Plasma (Cmax) at Cycle 4
Description: Maximum measured concentration of Ezabenlimab (BI 754091) at Cycle 4 in Part 2 (combination therapy) in plasma (Cmax) is reported.
Time Frame: Within 5 min before and at 1 h, 2h15min, 6h, 24h, 168h, 336h after dosing in Cycle 4. Also, Within 5 min before Cycle 5 dose.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram / milliliter (µg/mL)
Arm/Group | Part 2: 120 mg of BI 836880/ 240 mg Ezabenlimab | Part 2: 360 mg BI 836880/ 240 mg Ezabenlimab | Part 2: 720 mg BI 836880 / 240 mg Ezabenlimab
Number analyzed (Participants) | 2 | 2 | 3
microgram / milliliter (µg/mL) | 129 (13.8) | 106 (40.2) | 132 (37.9)

12. Secondary Outcome: Area Under the Concentration-time Curve of Ezabenlimab (BI 754091) in Part 2 in Plasma Over the Time Interval From 0 to 504 Hours (AUC0-504h) at Cycle 4
Description: as for outcome 10
Time Frame: as for outcome 11
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram/milliliter (h*µg/mL)
Arm/Group | Part 2: 120 mg of BI 836880/ 240 mg Ezabenlimab | Part 2: 360 mg BI 836880/ 240 mg Ezabenlimab | Part 2: 720 mg BI 836880 / 240 mg Ezabenlimab
Number analyzed (Participants) | 2 | 2 | 3
hour*microgram/milliliter (h*µg/mL) | 32200 (12.7) | 22900 (46.0) | 27600 (27.1)

ADVERSE EVENTS:
Time Frame: Part I: from first dose till last dose + 42 days, up to 444 + 42 days. Part II: from first dose till last dose + 42 days, up to 672 + 42 days.
Description: Treated set (TS) in monotherapy and in combination therapy: This patient set included all patients enrolled in the trial who were documented to have administrated at least one dose of BI 836880 monotherapy or BI 836880 and ezabenlimab (BI 754091) combination therapy.
Arm/Group | Part 1: 360 mg BI 836880 | Part 1: 720 mg BI 836880 | Part 2: 120 mg of BI 836880/ 240 mg Ezabenlimab | Part 2: 360 mg BI 836880/ 240 mg Ezabenlimab | Part 2: 720 mg BI 836880 / 240 mg Ezabenlimab
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/3 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 1/3 | 1/3 | 3/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: 360 mg BI 836880 (N=3) | Part 1: 720 mg BI 836880 (N=6) | Part 2: 120 mg of BI 836880/ 240 mg Ezabenlimab (N=3) | Part 2: 360 mg BI 836880/ 240 mg Ezabenlimab (N=3) | Part 2: 720 mg BI 836880 / 240 mg Ezabenlimab (N=6)
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Central nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: 360 mg BI 836880 (N=3) | Part 1: 720 mg BI 836880 (N=6) | Part 2: 120 mg of BI 836880/ 240 mg Ezabenlimab (N=3) | Part 2: 360 mg BI 836880/ 240 mg Ezabenlimab (N=3) | Part 2: 720 mg BI 836880 / 240 mg Ezabenlimab (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Visual field defect (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 3
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 1 | 1 | 1
Oedema (General disorders) | 0 | 1 | 0 | 1 | 2
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 2
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 1 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Osteoradionecrosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 2 | 1 | 1 | 1
Penile oedema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 2 | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT03972150/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT03972150/SAP_001.pdf